CLINICAL TRIAL: NCT07382362
Title: Strategies for the Prevention of Perioperative Neurological Complications in Cardiac Valve Surgery
Brief Title: Preventing Neurologic Complications in Valve Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-2452
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Left Atrial Appendage Closure
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Valve surgery with concomitant LAA suture closure: Concomitant suture closure of the LAA performed during surgical valve surgery.
  Interventions: Procedure: Left Atrial Appendage (LAA) Suture Closure
- Valve surgery alone (no LAA procedure): Standard surgical valve surgery without concomitant LAA suture closure.
  Interventions: Procedure: Surgical Valve Surgery

INTERVENTIONS:
Procedure: Left Atrial Appendage (LAA) Suture Closure — Concomitant suture closure of the LAA performed at the time of surgical valve surgery, at the discretion of the operating surgeon.
  Groups: Valve surgery with concomitant LAA suture closure
Procedure: Surgical Valve Surgery — Standard surgical valve repair or replacement performed according to routine clinical practice.
  Groups: Valve surgery alone (no LAA procedure)

SUMMARY:
In patients with valvular heart disease and atrial fibrillation (AF) undergoing surgical valve surgery, current guidelines recommend concomitant surgical management of the left atrial appendage (LAA) to prevent postoperative thromboembolic events, particularly neurologic embolic events. However, whether concomitant LAA management benefits patients without AF by reducing postoperative neurologic complications remains controversial.

Given these uncertainties, this study aims to evaluate whether concomitant LAA suture closure during surgical valve surgery is associated with a lower incidence of perioperative silent cerebral infarction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) without atrial fibrillation who are scheduled to undergo open (direct-vision) surgical heart valve surgery and who are informed about the study and provide written informed consent to participate.

Exclusion Criteria:

* History of prior cardiac surgery
* history of cerebral infarction (ischemic stroke)
* emergency surgery
* infective endocarditis
* pregnancy
* refusal or inability to provide informed consent/declines participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multicenter observational study conducted at four participating hospitals in China. Adult patients (≥18 years) without atrial fibrillation who are scheduled to undergo elective open surgical heart valve surgery and provide informed consent will be enrolled. Participants will be grouped according to whether concomitant left atrial appendage (LAA) suture closure is performed during the index operation. The primary outcome is perioperative silent brain infarction (SBI) assessed by brain MRI at approximately postoperative day 5. Secondary outcomes include stroke, myocardial infarction, all-cause death, cardiovascular death, and MACCE within 30 days after surgery, as well as SBI and MACCE (including rehospitalization for heart failure) within 1 year after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-27 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Silent brain infarction (SBI) | Approximately postoperative day 5
  Occurrence of SBI assessed by postoperative brain magnetic resonance imaging (MRI) performed at approximately postoperative day 5.

SECONDARY OUTCOMES:
Perioperative stroke | Within 30 days after surgery
  Incidence of clinically overt stroke within 30 days after surgery.
Perioperative all-cause mortality | Within 30 days after surgery
  Death from any cause within 30 days after surgery.
Perioperative MACCE | Within 30 days after surgery
  Incidence of major adverse cardiovascular and cerebrovascular events (MACCE), defined as a composite of stroke, myocardial infarction, all-cause death, or cardiovascular death occurring within 30 days after surgery.
Silent brain infarction (SBI) at 1 year | Occurrence of SBI assessed by brain MRI at 1 year after surgery.
  1 year after surgery
MACCE at 1 year | Within 1 year after surgery
  Incidence of major adverse cardiovascular and cerebrovascular events (MACCE) within 1 year after surgery, defined as a composite of stroke, myocardial infarction, all-cause death, cardiovascular death, or rehospitalization for heart failure.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Fuwai Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University First Hospita, Beijing, Beijing Municipality
  - Qingdao Cardiovascular Hospital, Qingdao
  - Fuwai Hospital Chinese Academy of Medical Sciences, Shenzhen, Shenzhen

IPD SHARING:
Plan to Share IPD: No